CLINICAL TRIAL: NCT05974059
Title: Single-arm, Open-label, Single-center Phase II Clinical Study of Cadonilimab Combined With CapeOX Regimen in Perioperative Treatment of Resectable Locally Advanced Gastric Cancer
Brief Title: Cadonilimab Combined With CapeOX Regimen in Perioperative Treatment of Resectable Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-N1-0036
Record Dates: First submitted 2023-07-24; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Locally Advanced Unresectable Gastric Adenocarcinoma
Keywords: Resectable locally advanced adenocarcinoma of the gastro-esophageal junction
MeSH Terms: interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab (Experimental): 10 mg/kg, d1, Q3W;
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Cadonilimab

INTERVENTIONS:
Drug: Oxaliplatin — Preoperative treatment：130mg/m2，iv, 2h，d1，Q3W; Postoperative treatment：130mg/m2，iv, 2h，d1，Q3W;
Drug: Capecitabine — Preoperative treatment：1000 mg /m2, PO，bid d1-14，Q3W； Postoperative treatment：1000 mg /m2, PO，bid. d1-14，Q3W；
Drug: Cadonilimab — Cadonilimab 10 mg/kg, d1, Q3W

SUMMARY:
The efficacy and safety of combination with Cadonilimab and CapeOX Regimen for neoadjuvant treatment of resectable locally advanced adenocarcinoma of the gastro-esophageal junction.

DETAILED DESCRIPTION:
This study was a single arm, open-label, single-center clinical study to evaluate the efficacy and safety of combination with Cadonilimab and CapeOX Regimen for neoadjuvant treatment of resectable locally advanced adenocarcinoma of the gastro-esophageal junction.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years ≤ age ≤ 75 years;
2. ECOG score 0-1;
3. Histologically confirmed gastric adenocarcinoma or adenocarcinoma of the gastroesophageal junction.
4. c stageII, III(T1-4a/N+ M0, T3-4a/N-M0, AJCC 8th edition of gastric cancer cTNM stage) were performed according to enhanced CT/MRI examination (combined with ultrasonic gastroscopy and diagnostic laparoscopy if necessary).
5. The study site and the operator can complete radical dissection of D2 lymph nodes (the number of examined lymph nodes must be at least 15 to ensure the operation quality), and R0 resection;
6. Physical condition and organ function allow for larger abdominal surgery;
7. It has adequate organ and bone marrow functions and is defined as follows:

1)Blood routine test: absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count(PLT)≥100×109/L; Hemoglobin (HGB)≥9.0 g/dL; 2)Liver function: Total serum bilirubin (TBIL) ≤1.5×upper limit of normal (ULN) is required for patients without liver metastasis. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5*ULN; 3)Renal function: creatinine clearance rate (Ccr)≥50 mL/min (calculated by Cockcroft/Gault formula); a Female: Ccr= (140-years) x Body Weight (kg) x 0.85 72 x serum creatinine (mg/dL) b Males: Ccr= (140-years) x Weight (kg) x 1.00 72 x serum creatinine (mg/dL) 4) Adequate coagulation, defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN; If the subject is receiving anticoagulant therapy, as long as the PT is within the intended range of the anticoagulant; 8 Left ventricular ejection fraction (LVEF)≥50% confirmed by echocardiography; 9 Agree and be able to comply with the protocol during the study; 10 Provide written informed consent prior to entering study screening and the patient is aware that she can withdraw from the study at any time during the study without loss; 11 Consent to provide blood and histological specimens

- Exclusion Criteria

1. Complication of upper gastrointestinal tract obstruction/hemorrhage or digestive dysfunction or malabsorption syndrome;
2. Concomitant severe uncontrolled concurrent infection or other serious uncontrolled concomitant disease, moderate or severe renal injury;
3. Prior anti-tumor therapy, including chemotherapy, radiotherapy, targeted therapy or immunotherapy;
4. Other malignancies (except basal or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ or breast cancer) in the past 5 years;
5. Uncontrolled pleural effusion, pericardial effusion or ascites;
6. Serious cardiovascular disease such as symptomatic coronary heart disease, congestive heart failure ≥Grade II, uncontrolled arrhythmia, myocardial infarction within 12 months prior to enrollment;
7. Allergic reaction to the drugs used in this study;
8. Use of steroids or other systemic immunosuppressive therapy 14 days prior to enrollment;
9. Patients receiving study medication within 4 weeks prior to enrollment (participating in other clinical trials);
10. Active autoimmune diseases;
11. Medical history of primary immunodeficiency;
12. Immunosuppressive medications were used within 4 weeks prior to the first dose of study treatment, excluding nasal spray, inhaled or other local corticosteroids or physiological doses of systemic corticosteroids (i.e. not more than 10 mg/day prednisone or equivalent dose of other corticosteroids), or the use of hormones to prevent contrast agent allergy;
13. Receiving an attenuated live vaccine within 4 weeks prior to the first dose of study treatment or scheduled for the duration of the study;
14. Known active tuberculosis;
15. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
16. HIV antibody positive, active hepatitis B or hepatitis C (HBV, HCV);
17. Pregnant or lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete remission rate (PCR) | up to 1 years
  Pathological complete response (pCR) rate is defined as the proportion of participants whose tumor in the stomach and lymph node completely disappeared, as determined by a pathologist.

SECONDARY OUTCOMES:
3-year disease-free survival rate of 3year (DFS) | up to 3 years
  3 years disease-free survival (DFS) rate is defined as proportion of participants who have no recurrence or metastasis after 3 years of radical treatment
Major pathological response rate (MPR) | up to 1 years
  Major pathological response (MPR) rate is defined as the proportion of participants whose percentage of residual tumor in the stomach and lymph node decreased to < 10%, as determined by a pathologist
Objective response rate(ORR) | up to 3 years
  Overall response rate ( ORR) is defined as proportion of participants who have a best response of CR or PR
Disease Control Rate (DCR) | up to 3 years
  Disease Control Rate (DCR) is defined as proportion of participants who have a best response of CR#PR or SD
Adverse Events（AEs） | up to 3 years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xuewei Ding, MD, Study Director — Tianjin Cancer Hospital Airport Hospital
Locations (1):
- Xuewei Ding, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No